CLINICAL TRIAL: NCT03769194
Title: Immunogenicity and Safety Study of VLA15, A Multivalent Recombinant OspA (Outer Surface Protein A) Based Vaccine Candidate Against Lyme Borreliosis, in Healthy Adults Aged 18 to 65 Years. A Randomized, Controlled, Observer-blind Phase 2 Study.
Brief Title: Immunogenicity and Safety Study of a Vaccine Against Lyme Borreliosis, in Healthy Adults Aged 18 to 65 Years. Randomized, Controlled, Observer-blind Phase 2 Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA15-201
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Lyme Borreliosis
Keywords: VLA15, Lyme Borreliosis, Vaccine
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VLA15 low dose (Active Comparator): VLA15 low dose with Alum.
  Interventions: Biological: VLA15
- VLA15 medium dose (Active Comparator): VLA15 medium dose with Alum.
  Interventions: Biological: VLA15
- VLA15 high dose (Active Comparator): VLA15 high dose with Alum.
  Interventions: Biological: VLA15
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA15 — a multivalent recombinant Outer surface protein A (OspA) based vaccine candidate
  Arms: VLA15 high dose; VLA15 low dose; VLA15 medium dose
Biological: Placebo — Placebo: PBS (Phosphate Buffered Saline)
  Arms: Placebo

SUMMARY:
This is a randomized, observer-blind, placebo controlled, multicenter Phase 2 study conducted in two study phases: a run-in phase and a main study phase. The study was investigated 3 doses of a multivalent OspA (Outer Surface Protein A) based Lyme vaccine (VLA15) in healthy adults aged 18 to 65 years of age. Study participants received 3 immunizations of the vaccine at a monthly interval. The study assessed the immune response as well as the safety profile of the vaccine.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, placebo controlled, multicenter Phase 2 study.

In the Run-in phase, a total of 120 subjects aged 18 to 40 years were randomized 1:1:1:1 to receive one of three VLA15 doses (VLA15 low dose (90 µg), VLA15 medium dose (135 µg), VLA15 high dose (180 µg)) or Placebo as intramuscular vaccinations on Days 1, 29 and 57.

Dosing was adjusted by injection volume.

In the Main Study phase, a total of 452 subjects aged 18 to 65 years were randomized 2:2:1 to receive VLA15 135 µg or VLA15 180 µg, the two dose groups were selected from the Run-in-Phase or placebo, as intramuscular vaccinations on Days 1, 29 and 57. Subjects were enrolled in two age groups (18-49 years and 50-65 years) in a ratio of approx. 2:1.

In both study phases, target was to enroll approx. 10 % or more of subjects that were baseline seropositive for Borrelia burgdorferi sensu latu (Bb s.l.).

ELIGIBILITY:
Inclusion Criteria:

Run-in phase:

1. Subject is aged 18 to 40 years at the day of screening (Visit 0);

Main Study phase:

1. Subject is aged18 to 65 years at the day of screening (Visit 0);

   Run-in phase and Main Study phase:
2. Subject is of good general health, including subjects with pharmacologically controlled chronic conditions;
3. Subject has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures;
4. If subject is of childbearing potential:

   1. Subject has a negative serum pregnancy test at screening (Visit 0);
   2. Subject agrees to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

1. Subject has a chronic illness related to Lyme borreliosis (LB), an active symptomatic LB (Lyme borreliosis) as suspected or diagnosed by a physician, or received treatment for LB (Lyme borreliosis) within the last 3 months prior to Visit 0;
2. Subject received previous vaccination against Lyme borreliosis (LB).;
3. Subject had a tick bite within 4 weeks prior to Visit 1;
4. Subject has a medical history of or currently has a clinically relevant disease (cardiovascular, respiratory, neurologic, psychiatric conditions) which poses a risk for participation in the study, based on investigators judgement, such as individuals with poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment. Subjects with pharmacologically controlled conditions like osteoarthritis, depression, or asthma are eligible;
5. Subject has a medical history of or currently has a neuroinflammatory or autoimmune disease, including Guillain Barré Syndrome;
6. Subject has a known thrombocytopenia, bleeding disorder, or received anticoagulants in the 3 weeks prior to first vaccination or until Day 57 (Visit 3), contraindicating intramuscular vaccination as judged by the investigator;
7. Subject has received an active or passive immunization within 28 days before first vaccination at Visit 1 and until Day 85; except for influenza (seasonal or pandemic) and pneumococcal vaccines which may be administered outside a 7-days interval before or after any trial vaccination;
8. Subject has received any other non-registered medicinal product in another clinical trial within 28 days prior to VLA15 vaccination at Visit 1 (Day 1) and throughout the entire study period or has received a registered medicinal product in another clinical trial within 28 days prior to VLA15 vaccination at Visit 1 (Day 1) and up to Day 85;
9. Subject has a known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired immunodeficiency, including infection with human immunodeficiency virus (HIV), status post organ transplantation or immuno-suppressive therapy within 30 days prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent 0.05 mg per kg/ per day. Topical and inhaled steroids are allowed;
10. Subject has a history of anaphylaxis or severe allergic reactions or a known hypersensitivity or allergic reactions to one of the components of the vaccine;
11. Subject had any malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled;
12. Subject had acute febrile infections within 10 days prior to first vaccination;
13. Subject is pregnant (positive serum pregnancy test at screening), has plans to become pregnant during the course of the study or is lactating at the time of enrollment. Women of childbearing potential that are unwilling or unable to employ an adequate birth control measure for the duration of the study.
14. Subject has donated blood or blood-derived products (plasma) within 30 days or received blood or blood-derived products (plasma) within 90 days prior to first vaccination in this study or plans to donate or use blood or blood products during the course of the study;
15. Subject has any condition that, in the opinion of the investigator, may compromise the subject's well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
16. Subject is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
17. Subject is in a dependent relationship with the sponsor, an investigator or other study team member, or the study center. Dependent relationships include close relatives and household members (i.e. children, partner/spouse, siblings, parents) as well as employees of the investigator or study center personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (6):
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Omega Medical Research, Warwick, Rhode Island
- Cevac Center for vaccinology, Ghent, Belgium
- Germany (2):
  - Berliner Centrum für Reise- und Tropenmedizin (BCRT), Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Derived] Bezay N, Wagner L, Kadlecek V, Obersriebnig M, Wressnigg N, Hochreiter R, Schneider M, Dubischar K, Derhaschnig U, Klingler A, Larcher-Senn J, Eder-Lingelbach S, Bender W. Optimisation of dose level and vaccination schedule for the VLA15 Lyme borreliosis vaccine candidate among healthy adults: two randomised, observer-blind, placebo-controlled, multicentre, phase 2 studies. Lancet Infect Dis. 2024 Sep;24(9):1045-1058. doi: 10.1016/S1473-3099(24)00175-0. Epub 2024 May 31. PMID 38830375

RESULTS

PARTICIPANT FLOW:
Groups:
- VLA15 Low Dose: VLA15 low dose with Alum.
  VLA15: a multivalent Outer surface protein A (OspA) based vaccine candidate
- VLA15 Medium Dose: VLA15 medium dose with Alum.
  VLA15: a multivalent Outer surface protein A (OspA) based vaccine candidate
- VLA15 High Dose: VLA15 high dose with Alum.
  VLA15: a multivalent Outer surface protein A (OspA) based vaccine candidate
Period: Overall Study
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Started | 29 | 214 | 205 | 124
Completed (Subjects that completed Day 85 (Visit 4)) | 25 | 196 | 197 | 115
Not Completed | 4 | 18 | 8 | 9
Not completed — Withdrawal by Subject | 0 | 7 | 4 | 1
Not completed — moved from study area | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 3 | 6 | 3 | 6
Not completed — other | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo | Total
Number analyzed (Participants) | 29 | 214 | 205 | 124 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.13) | 41.7 (13.26) | 41.6 (12.56) | 40.7 (12.80) | 40.8 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 117 | 108 | 71 | 312
  Male | 13 | 97 | 97 | 53 | 260
Race/Ethnicity, Customized [Number; unit: number of participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 2
  Black or African American | 4 | 3 | 6 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 25 | 208 | 196 | 120 | 549
  Other | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype ST1 to ST6
Description: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) against each OspA (Outer Surface Protein A) serotype ST1 to ST6, determined by ELISA at Day 85.
  GMTs are calculated based on the number of subjects with non-missing results.
Time Frame: at Day 85 / Month 3
Population: Overall Number of Participants Analyzed Per Protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 192 | 194 | 121
U/mL
  ST1 Day 85 | 74.3 [46.4 to 119.0] | 101.9 [87.1 to 119.4] | 115.8 [98.8 to 135.7] | 21.7 [20.0 to 23.6]
  ST2 Day 85 | 180.9 [124.8 to 262.3] | 279.3 [247.1 to 315.8] | 303.7 [266.5 to 346.1] | 21.1 [20.0 to 22.3]
  ST3 Day 85 | 267.4 [194.8 to 367.1] | 283.2 [248.2 to 323.1] | 308.6 [266.8 to 356.8] | 20.8 [19.8 to 21.8]
  ST4 Day 85 | 117.0 [76.6 to 178.7] | 170.9 [150.5 to 194.2] | 190.7 [165.9 to 219.2] | 21.8 [20.4 to 23.4]
  ST5 Day 85 | 118.3 [78.3 to 178.9] | 176.0 [154.2 to 201.0] | 199.6 [172.5 to 230.9] | 21.4 [20.2 to 22.6]
  ST6 Day 85 | 115.6 [76.5 to 174.7] | 183.6 [161.7 to 208.4] | 208.7 [181.8 to 239.6] | 21.8 [20.3 to 23.4]

2. Secondary Outcome: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6)
Description: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) against each OspA (Outer Surface Protein A) (Outer Surface Protein A) serotype (ST1 to ST6), determined by ELISA.
  GMTs are calculated based on the number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 192 | 194 | 121
U/mL
  ST1 Day 1 | 20.8 [19.2 to 22.5] | 20.5 [19.8 to 21.3] | 20.2 [19.8 to 20.6] | 21.6 [19.9 to 23.5]
  ST1 Day 29 | 21.1 [18.9 to 23.5] | 21.8 [20.0 to 23.8] | 21.2 [20.1 to 22.4] | 21.7 [20.0 to 23.7]
  ST1 Day 57 | 32.7 [25.1 to 42.6] | 37.5 [32.4 to 43.3] | 41.2 [35.7 to 47.5] | 21.9 [20.1 to 23.8]
  ST1 Day 180 | 26.2 [19.9 to 34.5] | 32.8 [28.8 to 37.3] | 33.9 [30.0 to 38.3] | 21.0 [19.8 to 22.3]
  ST1 Day 236 | 22.2 [18.8 to 26.1] | 25.7 [22.8 to 28.8] | 26.2 [23.1 to 29.7] | 21.5 [19.6 to 23.6]
  ST1 Day 365 | 20.9 [19.1 to 22.9] | 23.4 [21.4 to 25.6] | 23.0 [21.3 to 24.9] | 21.4 [19.9 to 22.9]
  ST2 Day 1 | 21.3 [18.7 to 24.2] | 20.0 [20.0 to 20.0] | 20.1 [19.9 to 20.2] | 20.7 [19.7 to 21.8]
  ST2 Day 29 | 21.1 [18.9 to 23.7] | 21.1 [20.0 to 22.2] | 21.4 [20.5 to 22.4] | 21.0 [19.9 to 22.1]
  ST2 Day 57 | 69.0 [47.7 to 99.8] | 89.2 [75.9 to 104.9] | 107.8 [92.7 to 125.2] | 21.3 [20.0 to 22.6]
  ST2 Day 180 | 41.2 [29.3 to 57.9] | 62.5 [54.5 to 71.7] | 67.1 [58.3 to 77.1] | 20.6 [19.7 to 21.5]
  ST2 Day 236 | 26.6 [21.2 to 33.4] | 36.8 [32.1 to 42.2] | 35.7 [30.9 to 41.2] | 20.5 [19.5 to 21.5]
  ST2 Day 365 | 21.8 [19.2 to 24.7] | 24.6 [22.8 to 26.6] | 24.8 [23.1 to 26.6] | 20.6 [19.7 to 21.5]
  ST3 Day 1 | 21.9 [19.1 to 25.1] | 20.4 [20.0 to 20.8] | 20.1 [19.9 to 20.4] | 20.4 [19.6 to 21.2]
  ST3 Day 29 | 23.7 [20.0 to 28.0] | 21.7 [20.2 to 23.2] | 21.2 [20.3 to 22.1] | 20.8 [19.8 to 21.9]
  ST3 Day 57 | 110.2 [71.1 to 171.0] | 123.8 [104.4 to 146.9] | 145.8 [122.8 to 173.0] | 21.2 [20.0 to 22.6]
  ST3 Day 180 | 53.1 [35.6 to 79.1] | 63.1 [55.2 to 72.2] | 68.7 [59.5 to 79.2] | 20.5 [19.8 to 21.3]
  ST3 Day 236 | 35.3 [25.7 to 48.6] | 35.8 [31.2 to 41.1] | 39.0 [33.3 to 45.8] | 20.6 [19.7 to 21.7]
  ST3 Day 365 | 25.2 [19.9 to 31.8] | 25.6 [23.5 to 27.9] | 27.0 [24.5 to 29.8] | 20.5 [19.8 to 21.3]
  ST4 Day 1 | 21.4 [18.7 to 24.4] | 21.0 [20.3 to 21.7] | 20.2 [19.9 to 20.6] | 21.7 [20.3 to 23.2]
  ST4 Day 29 | 22.1 [19.1 to 25.6] | 21.9 [20.4 to 23.6] | 21.4 [20.4 to 22.4] | 22.0 [20.4 to 23.6]
  ST4 Day 57 | 45.9 [32.8 to 64.2] | 57.4 [49.5 to 66.6] | 64.7 [55.5 to 75.5] | 22.0 [20.4 to 23.8]
  ST4 Day 180 | 32.8 [24.1 to 44.6] | 48.1 [42.5 to 54.5] | 49.3 [43.1 to 56.3] | 21.5 [20.2 to 22.9]
  ST4 Day 236 | 25.5 [20.6 to 31.5] | 32.8 [29.0 to 37.2] | 31.9 [27.7 to 36.6] | 21.7 [20.0 to 23.5]
  ST4 Day 365 | 21.8 [19.2 to 24.7] | 26.5 [24.2 to 28.9] | 25.5 [23.2 to 27.9] | 21.7 [20.3 to 23.2]
  ST5 Day 1 | 20.6 [19.4 to 21.8] | 20.7 [20.1 to 21.3] | 20.2 [19.8 to 20.5] | 21.4 [20.2 to 22.7]
  ST5 Day 29 | 20.7 [19.2 to 22.4] | 21.2 [20.0 to 22.5] | 21.0 [20.2 to 21.9] | 21.4 [20.1 to 22.7]
  ST5 Day 57 | 42.7 [29.8 to 61.3] | 57.9 [44.9 to 67.2] | 72.2 [61.6 to 84.7] | 21.5 [20.2 to 22.9]
  ST5 Day 180 | 26.7 [20.7 to 34.3] | 44.0 [38.8 to 49.8] | 50.0 [43.5 to 57.4] | 21.1 [20.0 to 22.3]
  ST5 Day 236 | 23.0 [19.6 to 27.0] | 31.0 [27.5 to 35.0] | 32.4 [28.0 to 37.4] | 21.5 [20.0 to 23.1]
  ST5 Day 365 | 21.7 [19.3 to 24.3] | 24.0 [22.3 to 25.8] | 24.9 [22.7 to 27.2] | 21.1 [20.0 to 22.2]
  ST6 Day 1 | 21.1 [18.9 to 23.5] | 21.3 [20.4 to 22.2] | 20.8 [20.1 to 21.6] | 21.6 [20.2 to 23.2]
  ST6 Day 29 | 21.1 [18.9 to 23.6] | 22.7 [21.2 to 24.3] | 22.0 [20.9 to 23.2] | 22.0 [20.4 to 23.7]
  ST6 Day 57 | 42.3 [29.8 to 60.1] | 55.5 [48.1 to 64.1] | 65.3 [55.6 to 76.7] | 22.1 [20.4 to 23.9]
  ST6 Day 180 | 30.1 [22.6 to 40.2] | 48.4 [42.8 to 54.8] | 51.4 [44.7 to 59.0] | 21.4 [20.1 to 22.8]
  ST6 Day 236 | 25.6 [20.7 to 31.8] | 33.4 [29.5 to 37.8] | 33.2 [28.6 to 38.6] | 22.1 [20.2 to 24.3]
  ST6 Day 365 | 22.1 [19.2 to 25.5] | 25.7 [23.8 to 27.9] | 26.0 [23.6 to 28.7] | 21.8 [20.3 to 23.3]

3. Secondary Outcome: SCRs (Seroconversion Rate) for Each OspA (Outer Surface Protein A) Serotype Specific IgG (Immunoglobulin G) (ST1 to ST6),
Description: Seroconversion for ELISA is defined as:
  * for subjects that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive (i.e. antibody titer of ≥40 U/mL) at a certain time point.
  * for subjects that are seropositive at Visit 1 (baseline): a ≥ 4-fold rise in IgG antibody titer from Visit 1.
  Percentages are based on the number of subjects with non-missing observations.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 192 | 194 | 121
percentage of subjects
  ST1 Day 29 | 0.0 [0.0 to 11.7] | 3.7 [1.8 to 7.4] | 3.1 [1.4 to 6.6] | 0.8 [0.1 to 4.6]
  ST1 Day 57 | 39.3 [23.6 to 57.6] | 37.2 [30.6 to 44.2] | 40.7 [34.1 to 47.8] | 1.7 [0.5 to 5.8]
  ST1 Day 180 | 11.5 [4.0 to 29.0] | 32.8 [26.4 to 39.9] | 35.4 [29.0 to 42.5] | 0.9 [0.2 to 4.8]
  ST1 Day 236 | 7.7 [2.1 to 24.1] | 17.2 [11.5 to 24.9] | 18.5 [12.5 to 26.4] | 2.6 [0.7 to 9.1]
  ST1 Day 365 | 4.0 [0.7 to 19.5] | 10.9 [7.2 to 16.3] | 8.9 [5.6 to 13.8] | 1.8 [0.5 to 6.2]
  ST2 Day 29 | 0.0 [0.0 to 11.7] | 2.6 [1.1 to 6.0] | 5.7 [3.2 to 9.9] | 0.8 [0.1 to 4.6]
  ST2 Day 57 | 67.9 [49.3 to 82.1] | 72.3 [65.5 to 78.1] | 79.9 [73.7 to 84.9] | 1.7 [0.5 to 5.8]
  ST2 Day 180 | 42.3 [25.5 to 61.1] | 66.1 [59.0 to 72.6] | 66.7 [59.7 to 73.0] | 0.9 [0.2 to 4.8]
  ST2 Day 236 | 19.2 [8.5 to 37.9] | 42.6 [34.2 to 51.5] | 38.7 [30.4 to 47.6] | 0.0 [0.0 to 4.8]
  ST2 Day 365 | 8.0 [2.2 to 25.0] | 15.3 [10.8 to 21.2] | 17.8 [13.0 to 23.8] | 0.9 [0.2 to 4.8]
  ST3 Day 29 | 6.9 [1.9 to 22.0] | 4.2 [2.1 to 8.0] | 3.6 [1.8 to 7.3] | 1.7 [0.5 to 5.9]
  ST3 Day 57 | 75.0 [56.6 to 87.3] | 80.1 [73.9 to 85.1] | 84.0 [78.2 to 88.5] | 2.5 [0.8 to 7.0]
  ST3 Day 180 | 50.0 [32.1 to 67.9] | 68.9 [61.8 to 75.1] | 69.3 [62.4 to 75.4] | 1.8 [0.5 to 6.2]
  ST3 Day 236 | 34.6 [19.4 to 53.8] | 39.3 [31.1 to 48.2] | 42.0 [33.5 to 51.0] | 2.6 [0.7 to 9.1]
  ST3 Day 365 | 12.0 [4.2 to 30.0] | 17.5 [12.7 to 23.6] | 19.9 [14.9 to 26.1] | 1.8 [0.5 to 6.2]
  ST4 Day 29 | 3.4 [0.6 to 17.2] | 2.6 [1.1 to 6.0] | 3.6 [1.8 to 7.3] | 0.8 [0.1 to 4.6]
  ST4 Day 57 | 50.0 [32.6 to 67.4] | 58.6 [51.6 to 65.4] | 67.0 [60.1 to 73.2] | 0.8 [0.1 to 4.5]
  ST4 Day 180 | 30.8 [16.5 to 50.0] | 57.4 [50.1 to 64.3] | 58.2 [51.1 to 65.0] | 0.9 [0.2 to 4.8]
  ST4 Day 236 | 15.4 [6.2 to 33.5] | 36.1 [28.1 to 44.9] | 31.9 [24.2 to 40.8] | 1.3 [0.2 to 7.1]
  ST4 Day 365 | 8.0 [2.2 to 25.0] | 19.7 [14.6 to 26.0] | 16.8 [12.1 to 22.7] | 2.7 [0.9 to 7.5]
  ST5 Day 29 | 0.0 [0.0 to 11.7] | 1.6 [0.5 to 4.5] | 2.6 [1.1 to 5.9] | 0.0 [0.0 to 3.1]
  ST5 Day 57 | 42.9 [26.5 to 60.9] | 58.1 [51.0 to 64.9] | 67.5 [60.7 to 73.7] | 0.0 [0.0 to 3.1]
  ST5 Day 180 | 19.2 [8.5 to 37.9] | 49.7 [42.6 to 56.9] | 55.0 [47.9 to 61.9] | 0.9 [0.2 to 4.8]
  ST5 Day 236 | 11.5 [4.0 to 29.0] | 32.0 [24.4 to 40.7] | 31.9 [24.2 to 40.8] | 1.3 [0.2 to 7.1]
  ST5 Day 365 | 8.0 [2.2 to 25.0] | 13.1 [9.0 to 18.8] | 13.1 [9.0 to 18.6] | 0.9 [0.2 to 4.8]
  ST6 Day 29 | 0.0 [0.0 to 11.7] | 6.3 [3.6 to 10.7] | 4.6 [2.5 to 8.6] | 1.7 [0.5 to 5.9]
  ST6 Day 57 | 42.9 [26.5 to 60.9] | 54.5 [47.4 to 61.4] | 60.3 [53.3 to 66.9] | 1.7 [0.5 to 5.8]
  ST6 Day 180 | 23.1 [11.0 to 42.1] | 54.1 [46.9 to 61.2] | 53.4 [46.3 to 60.4] | 2.6 [0.9 to 7.5]
  ST6 Day 236 | 15.4 [6.2 to 33.5] | 35.2 [27.3 to 44.1] | 31.1 [23.5 to 39.9] | 3.9 [1.4 to 11.0]
  ST6 Day 365 | 8.0 [2.2 to 25.0] | 16.9 [12.2 to 23.0] | 13.6 [9.5 to 19.2] | 3.5 [1.4 to 8.7]

4. Secondary Outcome: GMFR (Geometric Mean of the Fold Rise as Compared to Baseline) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6)
Description: GMFR (Geometric Mean of the Fold Rise as compared to baseline) for IgG (Immunoglobulin G) against each OspA (Outer Surface Protein A) serotype (ST1 to ST6), determined by ELISA.
  Calculations are based on number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean of the Fold Rise
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 192 | 194 | 121
Geometric Mean of the Fold Rise
  ST1 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST1 Day 57 | 1.6 [1.2 to 2.1] | 1.8 [1.6 to 2.1] | 2.0 [1.8 to 2.4] | 1.0 [1.0 to 1.0]
  ST1 Day 180 | 1.3 [1.0 to 1.6] | 1.6 [1.4 to 1.8] | 1.7 [1.5 to 1.9] | 1.0 [1.0 to 1.0]
  ST1 Day 236 | 1.1 [0.9 to 1.3] | 1.3 [1.1 to 1.4] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.1]
  ST1 Day 365 | 1.0 [0.9 to 1.1] | 1.1 [1.1 to 1.2] | 1.1 [1.1 to 1.2] | 1.0 [1.0 to 1.1]
  ST2 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 3.2 [2.2 to 4.7] | 4.5 [3.8 to 5.2] | 5.4 [4.6 to 6.2] | 1.0 [1.0 to 1.1]
  ST2 Day 180 | 1.9 [1.4 to 2.7] | 3.1 [2.7 to 3.6] | 3.3 [2.9 to 3.8] | 1.0 [1.0 to 1.0]
  ST2 Day 236 | 1.2 [1.0 to 1.6] | 1.8 [1.6 to 2.1] | 1.8 [1.5 to 2.1] | 1.0 [1.0 to 1.0]
  ST2 Day 365 | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3] | 1.0 [1.0 to 1.0]
  ST3 Day 29 | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.1]
  ST3 Day 57 | 5.0 [3.2 to 7.8] | 6.1 [5.1 to 7.2] | 7.2 [6.1 to 8.6] | 1.0 [1.0 to 1.1]
  ST3 Day 180 | 2.4 [1.6 to 3.6] | 3.1 [2.7 to 3.5] | 3.4 [3.0 to 3.9] | 1.0 [1.0 to 1.1]
  ST3 Day 236 | 1.6 [1.2 to 2.2] | 1.8 [1.5 to 2.0] | 1.9 [1.6 to 2.3] | 1.0 [1.0 to 1.1]
  ST3 Day 365 | 1.2 [1.0 to 1.4] | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.1]
  ST4 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST4 Day 57 | 2.1 [1.5 to 3.0] | 2.7 [2.4 to 3.2] | 3.2 [2.7 to 3.7] | 1.0 [1.0 to 1.0]
  ST4 Day 180 | 1.5 [1.1 to 2.1] | 2.3 [2.0 to 2.6] | 2.4 [2.1 to 2.8] | 1.0 [1.0 to 1.0]
  ST4 Day 236 | 1.2 [0.9 to 1.5] | 1.6 [1.4 to 1.8] | 1.6 [1.4 to 1.8] | 1.0 [1.0 to 1.1]
  ST4 Day 365 | 1.1 [1.0 to 1.2] | 1.3 [1.2 to 1.4] | 1.3 [1.1 to 1.4] | 1.0 [1.0 to 1.1]
  ST5 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 2.1 [1.5 to 3.0] | 2.8 [2.4 to 3.2] | 3.6 [3.1 to 4.2] | 1.0 [1.0 to 1.0]
  ST5 Day 180 | 1.3 [1.0 to 1.7] | 2.1 [1.9 to 2.4] | 2.5 [2.2 to 2.8] | 1.0 [1.0 to 1.0]
  ST5 Day 236 | 1.1 [0.9 to 1.3] | 1.5 [1.4 to 1.7] | 1.6 [1.4 to 1.8] | 1.0 [1.0 to 1.0]
  ST5 Day 365 | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.2] | 1.2 [1.1 to 1.3] | 1.0 [1.0 to 1.0]
  ST6 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST6 Day 57 | 2.0 [1.4 to 2.8] | 2.6 [2.3 to 3.0] | 3.1 [2.7 to 3.7] | 1.0 [1.0 to 1.0]
  ST6 Day 180 | 1.4 [1.1 to 1.9] | 2.3 [2.0 to 2.6] | 2.5 [2.1 to 2.8] | 1.0 [1.0 to 1.1]
  ST6 Day 236 | 1.2 [1.0 to 1.5] | 1.6 [1.4 to 1.8] | 1.6 [1.4 to 1.9] | 1.0 [1.0 to 1.1]
  ST6 Day 365 | 1.1 [1.0 to 1.3] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.4] | 1.0 [1.0 to 1.1]

5. Secondary Outcome: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 18 - 49 Years
Description: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) against each OspA (Outer Surface Protein A) serotype (ST1 to ST6), determined by ELISA, stratified by age group - Group 18 - 49 years.
  GMTs are calculated based on the number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 133 | 136 | 88
U/mL
  ST1 Day 1 | 20.8 [19.2 to 22.5] | 20.3 [19.7 to 21.0] | 20.3 [19.7 to 20.8] | 22.0 [19.6 to 24.6]
  ST1 Day 29 | 21.1 [18.9 to 23.5] | 20.9 [19.7 to 22.1] | 21.4 [19.9 to 23.0] | 22.0 [19.6 to 24.6]
  ST1 Day 57 | 32.7 [25.1 to 42.6] | 34.8 [30.0 to 40.3] | 43.6 [36.5 to 52.0] | 22.4 [19.9 to 25.2]
  ST1 Day 85 | 74.3 [46.4 to 119.0] | 105.2 [88.8 to 124.5] | 129.6 [107.6 to 156.2] | 21.9 [19.6 to 24.5]
  ST1 Day 180 | 26.2 [19.9 to 34.5] | 31.7 [27.5 to 36.4] | 34.7 [29.7 to 40.5] | 21.0 [19.5 to 22.7]
  ST1 Day 236 | 22.2 [18.8 to 26.1] | 26.1 [22.5 to 30.3] | 26.4 [22.4 to 31.2] | 21.7 [19.3 to 24.4]
  ST1 Day 365 | 20.9 [19.1 to 22.9] | 23.0 [21.1 to 25.1] | 23.8 [21.4 to 26.5] | 21.7 [19.7 to 23.9]
  ST2 Day 1 | 21.3 [18.7 to 24.2] | 20.0 [20.0 to 20.0] | 20.1 [19.9 to 20.3] | 21.0 [19.6 to 22.5]
  ST2 Day 29 | 21.1 [18.9 to 23.7] | 20.7 [19.9 to 21.5] | 21.4 [20.5 to 22.3] | 21.0 [19.6 to 22.4]
  ST2 Day 57 | 69.0 [47.7 to 99.8] | 89.5 [74.2 to 107.9] | 121.4 [102.4 to 143.9] | 21.4 [19.8 to 23.2]
  ST2 Day 85 | 180.9 [124.8 to 262.3] | 296.5 [258.6 to 339.9] | 322.1 [277.1 to 374.4] | 21.2 [19.8 to 22.7]
  ST2 Day 180 | 41.2 [29.3 to 57.9] | 64.5 [54.7 to 76.0] | 71.8 [60.8 to 84.7] | 20.5 [19.5 to 21.6]
  ST2 Day 236 | 26.6 [21.2 to 33.4] | 39.6 [33.5 to 46.8] | 37.0 [31.2 to 43.9] | 20.6 [19.4 to 22.0]
  ST2 Day 365 | 21.8 [19.2 to 24.7] | 24.5 [22.4 to 26.8] | 25.1 [23.0 to 27.4] | 20.5 [19.5 to 21.6]
  ST3 Day 1 | 21.9 [19.1 to 25.1] | 20.3 [19.9 to 20.7] | 20.2 [19.8 to 20.5] | 20.6 [19.5 to 21.7]
  ST3 Day 29 | 23.7 [20.0 to 28.0] | 21.0 [20.1 to 21.9] | 21.7 [20.5 to 23.0] | 20.7 [19.6 to 21.9]
  ST3 Day 57 | 110.2 [71.1 to 171.0] | 122.6 [101.3 to 148.3] | 159.4 [130.1 to 195.2] | 21.3 [19.7 to 22.9]
  ST3 Day 85 | 267.4 [194.8 to 367.1] | 295.1 [255.6 to 340.8] | 334.2 [282.1 to 395.9] | 20.7 [19.6 to 21.8]
  ST3 Day 180 | 53.1 [35.6 to 79.1] | 60.7 [51.7 to 71.2] | 73.0 [61.3 to 86.9] | 20.0 [20.0 to 20.0]
  ST3 Day 236 | 35.3 [25.7 to 48.6] | 35.8 [30.4 to 42.2] | 39.9 [33.0 to 48.3] | 20.2 [19.8 to 20.7]
  ST3 Day 365 | 25.2 [19.9 to 31.8] | 25.4 [23.2 to 27.8] | 28.0 [24.7 to 31.8] | 20.2 [19.8 to 20.7]
  ST4 Day 1 | 21.4 [18.7 to 24.4] | 20.8 [20.0 to 21.6] | 20.3 [19.9 to 20.8] | 22.0 [20.2 to 24.0]
  ST4 Day 29 | 22.1 [19.1 to 25.6] | 21.5 [20.4 to 22.8] | 21.5 [20.3 to 22.8] | 22.3 [20.4 to 24.4]
  ST4 Day 57 | 45.9 [32.8 to 64.2] | 56.9 [48.3 to 67.1] | 71.4 [59.1 to 86.3] | 22.4 [20.4 to 24.6]
  ST4 Day 85 | 117.0 [76.6 to 178.7] | 177.1 [154.5 to 203.1] | 206.8 [175.0 to 244.3] | 22.1 [20.3 to 24.1]
  ST4 Day 180 | 32.8 [24.1 to 44.6] | 48.2 [41.8 to 55.6] | 53.2 [44.9 to 63.0] | 21.7 [20.0 to 23.5]
  ST4 Day 236 | 25.5 [20.6 to 31.5] | 34.9 [29.9 to 40.8] | 33.6 [28.1 to 40.1] | 21.2 [19.5 to 23.2]
  ST4 Day 365 | 21.8 [19.2 to 24.7] | 26.7 [24.2 to 29.5] | 26.7 [23.5 to 30.3] | 21.4 [19.9 to 23.0]
  ST5 Day 1 | 20.6 [19.4 to 21.8] | 20.4 [19.9 to 20.9] | 20.2 [19.8 to 20.8] | 21.5 [20.0 to 23.1]
  ST5 Day 29 | 20.7 [19.2 to 22.4] | 20.6 [19.9 to 21.3] | 21.1 [20.1 to 22.1] | 21.4 [20.0 to 22.9]
  ST5 Day 57 | 42.7 [29.8 to 61.3] | 56.6 [47.8 to 67.0] | 80.7 [66.3 to 98.1] | 21.6 [20.0 to 23.3]
  ST5 Day 85 | 118.3 [78.3 to 178.9] | 180.7 [156.8 to 208.2] | 218.3 [183.6 to 259.7] | 21.4 [20.0 to 22.9]
  ST5 Day 180 | 26.7 [20.7 to 34.3] | 42.5 [36.7 to 49.1] | 54.6 [45.9 to 64.8] | 20.8 [19.7 to 21.9]
  ST5 Day 236 | 23.0 [19.6 to 27.0] | 31.9 [27.5 to 37.1] | 33.4 [27.7 to 40.2] | 21.0 [19.6 to 22.6]
  ST5 Day 365 | 21.7 [19.3 to 24.3] | 24.0 [22.2 to 26.0] | 26.0 [23.0 to 29.5] | 20.8 [19.7 to 21.9]
  ST6 Day 1 | 21.1 [18.9 to 23.5] | 20.8 [20.0 to 21.5] | 21.2 [20.1 to 22.4] | 21.7 [20.0 to 23.6]
  ST6 Day 29 | 21.1 [18.9 to 23.6] | 22.3 [21.0 to 23.7] | 22.2 [20.8 to 23.7] | 22.1 [20.3 to 24.0]
  ST6 Day 57 | 42.3 [29.8 to 60.1] | 54.5 [46.2 to 64.3] | 72.3 [59.2 to 88.3] | 22.3 [20.3 to 24.4]
  ST6 Day 85 | 115.6 [76.5 to 174.7] | 185.8 [162.2 to 213.0] | 225.6 [191.9 to 265.3] | 21.8 [20.1 to 23.7]
  ST6 Day 180 | 30.1 [22.6 to 40.2] | 46.7 [40.4 to 53.9] | 54.2 [45.5 to 64.4] | 20.6 [19.7 to 21.4]
  ST6 Day 236 | 25.6 [20.7 to 31.8] | 34.6 [29.8 to 40.2] | 34.6 [28.7 to 41.9] | 21.4 [19.7 to 23.2]
  ST6 Day 365 | 22.1 [19.2 to 25.5] | 25.5 [23.3 to 27.9] | 27.7 [24.3 to 31.6] | 21.4 [20.1 to 22.7]

6. Secondary Outcome: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 50 - 65 Years
Description: GMTs (Geometric Mean Titers) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6), determined by ELISA, stratified by age group - Group 50 - 65 years.
  GMTs are calculated based on the number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Population: In the elderly age group no participants were included in the VLA15 low dose, that's the reason why the number of participants is zero.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 0 | 59 | 58 | 33
U/mL
  ST1 Day 1 |  | 21.0 [19.0 to 23.3] | 20.0 [20.0 to 20.0] | 20.6 [19.4 to 22.0]
  ST1 Day 29 |  | 24.2 [18.7 to 31.4] | 20.9 [19.5 to 22.5] | 21.0 [19.6 to 22.6]
  ST1 Day 57 |  | 44.5 [31.7 to 62.3] | 36.2 [28.6 to 45.8] | 20.5 [19.5 to 21.6]
  ST1 Day 85 |  | 95.3 [67.2 to 135.1] | 89.2 [66.0 to 120.4] | 21.2 [19.5 to 23.1]
  ST1 Day 180 |  | 35.4 [26.8 to 46.9] | 32.1 [26.4 to 39.0] | 21.0 [19.6 to 22.5]
  ST1 Day 236 |  | 24.5 [20.4 to 29.4] | 25.6 [21.4 to 30.5] | 20.9 [19.1 to 22.9]
  ST1 Day 365 |  | 24.3 [19.6 to 30.1] | 21.4 [19.6 to 23.2] | 20.5 [19.4 to 21.7]
  ST2 Day 1 |  | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST2 Day 29 |  | 22.0 [18.9 to 25.7] | 21.6 [19.4 to 24.0] | 20.9 [19.1 to 22.8]
  ST2 Day 57 |  | 88.7 [64.1 to 122.5] | 81.5 [60.4 to 110.2] | 20.9 [19.1 to 22.8]
  ST2 Day 85 |  | 245.5 [190.3 to 316.6] | 265.0 [204.2 to 344.0] | 20.8 [19.2 to 22.4]
  ST2 Day 180 |  | 58.5 [45.4 to 75.3] | 57.4 [44.1 to 74.5] | 20.8 [19.2 to 22.4]
  ST2 Day 236 |  | 30.5 [24.1 to 38.7] | 32.7 [24.8 to 43.1] | 20.0 [20.0 to 20.0]
  ST2 Day 365 |  | 24.9 [21.3 to 29.2] | 24.1 [21.3 to 27.3] | 20.9 [19.1 to 22.7]
  ST3 Day 1 |  | 20.7 [19.7 to 21.7] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  ST3 Day 29 |  | 23.3 [18.9 to 28.7] | 20.0 [20.0 to 20.0] | 21.2 [18.8 to 23.8]
  ST3 Day 57 |  | 126.7 [88.0 to 182.4] | 118.3 [85.7 to 163.1] | 21.1 [18.9 to 23.6]
  ST3 Day 85 |  | 258.9 [194.9 to 343.8] | 256.5 [193.5 to 340.0] | 21.1 [19.0 to 23.4]
  ST3 Day 180 |  | 68.8 [53.5 to 88.4] | 59.7 [46.4 to 76.7] | 21.9 [19.1 to 25.0]
  ST3 Day 236 |  | 35.7 [27.3 to 46.8] | 36.9 [27.2 to 50.1] | 22.0 [18.0 to 26.9]
  ST3 Day 365 |  | 26.0 [21.5 to 31.5] | 24.8 [21.6 to 28.4] | 21.3 [18.7 to 24.2]
  ST4 Day 1 |  | 21.3 [19.8 to 23.0] | 20.0 [20.0 to 20.0] | 20.9 [19.1 to 22.9]
  ST4 Day 29 |  | 22.9 [18.7 to 28.0] | 21.0 [19.4 to 22.8] | 21.2 [18.8 to 23.8]
  ST4 Day 57 |  | 58.6 [42.6 to 80.6] | 51.4 [39.8 to 66.4] | 21.2 [18.8 to 23.9]
  ST4 Day 85 |  | 158.2 [119.5 to 209.4] | 158.1 [122.5 to 203.9] | 21.1 [18.9 to 23.4]
  ST4 Day 180 |  | 48.0 [37.5 to 61.5] | 41.3 [33.6 to 50.9] | 21.1 [18.9 to 23.6]
  ST4 Day 236 |  | 28.0 [23.1 to 33.8] | 28.0 [22.7 to 34.7] | 23.1 [18.7 to 28.5]
  ST4 Day 365 |  | 26.0 [21.7 to 31.1] | 22.9 [20.9 to 25.1] | 22.5 [19.4 to 26.1]
  ST5 Day 1 |  | 21.4 [19.8 to 23.0] | 20.0 [20.0 to 20.0] | 21.0 [19.0 to 23.4]
  ST5 Day 29 |  | 22.7 [19.0 to 27.1] | 20.8 [19.2 to 22.6] | 21.3 [18.7 to 24.3]
  ST5 Day 57 |  | 61.0 [44.9 to 82.9] | 55.7 [42.5 to 72.8] | 21.3 [18.7 to 24.2]
  ST5 Day 85 |  | 166.4 [124.1 to 223.0] | 162.1 [124.0 to 211.9] | 21.2 [18.8 to 23.9]
  ST5 Day 180 |  | 47.4 [37.2 to 60.5] | 40.8 [32.6 to 51.1] | 21.9 [19.1 to 25.2]
  ST5 Day 236 |  | 28.8 [23.4 to 35.6] | 30.2 [24.1 to 37.7] | 23.1 [18.6 to 28.7]
  ST5 Day 365 |  | 23.9 [20.5 to 27.8] | 22.4 [20.2 to 24.7] | 21.9 [19.1 to 25.2]
  ST6 Day 1 |  | 22.6 [20.3 to 25.1] | 20.0 [20.0 to 20.0] | 21.4 [18.7 to 24.4]
  ST6 Day 29 |  | 23.6 [19.9 to 28.1] | 21.6 [19.6 to 23.9] | 21.7 [18.3 to 25.8]
  ST6 Day 57 |  | 58.0 [43.2 to 77.7] | 51.4 [39.3 to 67.1] | 21.7 [18.4 to 25.6]
  ST6 Day 85 |  | 178.7 [136.2 to 236.3] | 174.3 [133.9 to 226.9] | 21.6 [18.5 to 25.3]
  ST6 Day 180 |  | 52.3 [41.1 to 66.5] | 45.5 [36.1 to 57.3] | 23.6 [19.2 to 28.8]
  ST6 Day 236 |  | 30.3 [24.1 to 38.1] | 30.1 [23.6 to 38.3] | 24.6 [18.0 to 33.6]
  ST6 Day 365 |  | 26.2 [22.2 to 30.9] | 22.5 [20.2 to 25.0] | 22.8 [18.7 to 27.8]

7. Secondary Outcome: SCRs (Seroconversion Rate) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 18 - 49 Years
Description: SCRs (Seroconversion Rate) for Seroconversion for ELISA is defined as:
  * for subjects that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive (i.e. antibody titer of ≥40 U/mL) at a vertain time point.
  * for subjects that are seropositive at Visit 1 (baseline): a ≥ 4-fold rise in IgG antibody titer from Visit 1.
  Percentages are based on the number of subjects with non-missing observations.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 133 | 136 | 88
percentage of subjects
  ST1 Day 29 | 0.0 [0.0 to 11.7] | 2.3 [0.8 to 6.4] | 2.9 [1.1 to 7.3] | 0.0 [0.0 to 4.2]
  ST1 Day 57 | 39.3 [23.6 to 57.6] | 36.1 [28.4 to 44.5] | 43.4 [35.3 to 51.8] | 1.1 [0.2 to 6.2]
  ST1 Day 85 | 65.4 [46.2 to 80.6] | 85.9 [78.9 to 90.9] | 85.6 [78.6 to 90.6] | 0.0 [0.0 to 4.3]
  ST1 Day 180 | 11.5 [4.0 to 29.0] | 31.2 [23.7 to 39.8] | 36.4 [28.7 to 44.8] | 0.0 [0.0 to 4.5]
  ST1 Day 236 | 7.7 [2.1 to 24.1] | 18.2 [11.5 to 27.5] | 17.9 [11.1 to 27.4] | 1.7 [0.3 to 9.1]
  ST1 Day 365 | 4.0 [0.7 to 19.5] | 11.3 [6.8 to 18.1] | 10.5 [6.4 to 16.9] | 1.2 [0.2 to 6.6]
  ST2 Day 29 | 0.0 [0.0 to 11.7] | 2.3 [0.8 to 6.4] | 6.6 [3.5 to 12.1] | 0.0 [0.0 to 4.2]
  ST2 Day 57 | 67.9 [49.3 to 82.1] | 72.9 [64.8 to 79.8] | 85.3 [78.4 to 90.3] | 1.1 [0.2 to 6.2]
  ST2 Day 85 | 88.5 [71.0 to 96.0] | 100 [97.1 to 100] | 96.2 [91.4 to 98.4] | 1.2 [0.2 to 6.4]
  ST2 Day 180 | 42.3 [25.5 to 61.1] | 68.0 [59.4 to 75.5] | 69.7 [61.4 to 76.9] | 0.0 [0.0 to 4.5]
  ST2 Day 236 | 19.2 [8.5 to 37.9] | 47.7 [37.6 to 58.0] | 41.7 [31.7 to 52.3] | 0.0 [0.0 to 6.2]
  ST2 Day 365 | 8.0 [2.2 to 25.0] | 15.3 [10.0 to 22.7] | 18.8 [13.1 to 26.3] | 0.0 [0.0 to 4.5]
  ST3 Day 29 | 6.9 [1.9 to 22.0] | 3.0 [1.2 to 7.5] | 5.1 [2.5 to 10.2] | 1.1 [0.2 to 6.2]
  ST3 Day 57 | 75.0 [56.6 to 87.3] | 81.2 [73.7 to 86.9] | 85.3 [78.4 to 90.3] | 2.3 [0.6 to 7.9]
  ST3 Day 85 | 96.2 [81.1 to 99.3] | 98.4 [94.5 to 99.6] | 97.0 [92.5 to 98.8] | 1.2 [0.2 to 6.4]
  ST3 Day 180 | 50.0 [32.1 to 67.9] | 66.4 [57.7 to 74.1] | 70.5 [62.2 to 77.6] | 0.0 [0.0 to 4.5]
  ST3 Day 236 | 34.6 [19.4 to 53.8] | 39.8 [30.2 to 50.2] | 44.0 [33.9 to 54.7] | 1.7 [0.3 to 9.1]
  ST3 Day 365 | 12.0 [4.2 to 30.0] | 19.4 [13.4 to 27.2] | 21.8 [15.6 to 29.6] | 1.2 [0.2 to 6.6]
  ST4 Day 29 | 3.4 [0.6 to 17.2] | 2.3 [0.8 to 6.5] | 3.7 [1.6 to 8.3] | 1.1 [0.2 to 6.2]
  ST4 Day 57 | 50.0 [32.6 to 67.4] | 60.2 [51.7 to 68.1] | 71.3 [63.2 to 78.3] | 1.1 [0.2 to 6.2]
  ST4 Day 85 | 80.8 [62.1 to 91.5] | 96.1 [91.2 to 98.3] | 94.7 [89.5 to 97.4] | 1.2 [0.2 to 6.4]
  ST4 Day 180 | 30.8 [16.5 to 50.0] | 58.4 [49.6 to 66.7] | 60.6 [52.1 to 68.5] | 1.2 [0.2 to 6.6]
  ST4 Day 236 | 15.4 [6.2 to 33.5] | 38.6 [29.1 to 49.1] | 34.5 [25.2 to 45.2] | 0.0 [0.0 to 6.2]
  ST4 Day 365 | 8.0 [2.2 to 25.0] | 21.0 [14.7 to 29.0] | 18.0 [12.4 to 25.4] | 1.2 [0.2 to 6.6]
  ST5 Day 29 | 0.0 [0.0 to 11.7] | 0.8 [0.1 to 4.1] | 2.9 [1.1 to 7.3] | 0.0 [0.0 to 4.2]
  ST5 Day 57 | 42.9 [26.5 to 60.9] | 59.4 [50.9 to 67.4] | 72.8 [64.8 to 79.6] | 0.0 [0.0 to 4.2]
  ST5 Day 85 | 80.8 [62.1 to 91.5] | 94.5 [89.1 to 97.3] | 91.7 [85.7 to 95.3] | 0.0 [0.0 to 4.3]
  ST5 Day 180 | 19.2 [8.5 to 37.9] | 48.8 [40.2 to 57.5] | 59.1 [50.6 to 67.1] | 0.0 [0.0 to 4.5]
  ST5 Day 236 | 11.5 [4.0 to 29.0] | 33.0 [24.0 to 43.3] | 32.1 [23.1 to 42.7] | 0.0 [0.0 to 6.2]
  ST5 Day 365 | 8.0 [2.2 to 25.0] | 15.3 [10.0 to 22.7] | 15.0 [10.0 to 22.1] | 0.0 [0.0 to 4.5]
  ST6 Day 29 | 0.0 [0.0 to 11.7] | 6.8 [3.6 to 12.4] | 4.4 [2.0 to 9.3] | 2.3 [0.6 to 7.9]
  ST6 Day 57 | 42.9 [26.5 to 60.9] | 55.6 [47.2 to 63.8] | 64.0 [55.6 to 71.6] | 2.3 [0.6 to 7.9]
  ST6 Day 85 | 80.8 [62.1 to 91.5] | 95.3 [90.2 to 97.8] | 92.4 [86.6 to 95.8] | 1.2 [0.2 to 6.4]
  ST6 Day 180 | 23.1 [11.0 to 42.1] | 54.4 [45.7 to 62.9] | 53.8 [45.3 to 62.1] | 1.2 [0.2 to 6.6]
  ST6 Day 236 | 15.4 [6.2 to 33.5] | 38.6 [29.1 to 49.1] | 32.1 [23.1 to 42.7] | 3.4 [1.0 to 11.7]
  ST6 Day 365 | 8.0 [2.2 to 25.0] | 17.7 [12.0 to 25.4] | 15.8 [10.6 to 22.9] | 3.7 [1.3 to 10.2]

8. Secondary Outcome: SCRs (Seroconversion Rate) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 50 - 65 Years
Description: Seroconversion for ELISA is defined as:
  * for subjects that are seronegative at Visit 1 (baseline): a change from seronegative at Visit 1 to seropositive (i.e. antibody titer of ≥40 U/mL) at a vertain time point.
  * for subjects that are seropositive at Visit 1 (baseline): a ≥ 4-fold rise in IgG antibody titer from Visit 1.
  Percentages are based on the number of subjects with non-missing observations.
Time Frame: up to Day 365 / Month 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 0 | 59 | 58 | 33
percentage of subjects
  ST1 Day 29 |  | 6.9 [2.7 to 16.4] | 3.4 [1.0 to 11.7] | 3.1 [0.6 to 15.7]
  ST1 Day 57 |  | 39.7 [28.1 to 52.5] | 34.5 [23.6 to 47.3] | 3.0 [0.5 to 15.3]
  ST1 Day 85 |  | 71.2 [58.6 to 81.2] | 71.9 [59.2 to 81.9] | 3.0 [0.5 to 15.3]
  ST1 Day 180 |  | 36.2 [25.1 to 49.1] | 33.3 [22.5 to 46.3] | 3.1 [0.6 to 15.7]
  ST1 Day 236 |  | 14.7 [6.4 to 30.1] | 20.0 [10.0 to 35.9] | 5.6 [1.0 to 25.8]
  ST1 Day 365 |  | 10.2 [4.7 to 20.5] | 5.2 [1.8 to 14.1] | 3.2 [0.6 to 16.2]
  ST2 Day 29 |  | 3.4 [1.0 to 11.7] | 3.4 [1.0 to 11.7] | 3.1 [0.6 to 15.7]
  ST2 Day 57 |  | 70.7 [58.0 to 80.8] | 67.2 [54.4 to 77.9] | 3.0 [0.5 to 15.3]
  ST2 Day 85 |  | 94.9 [86.1 to 98.3] | 93.0 [83.3 to 97.2] | 3.0 [0.5 to 15.3]
  ST2 Day 180 |  | 62.1 [49.2 to 73.4] | 59.6 [46.7 to 71.4] | 3.1 [0.6 to 15.7]
  ST2 Day 236 |  | 29.4 [16.8 to 46.2] | 31.4 [18.6 to 48.0] | 0.0 [0.0 to 17.6]
  ST2 Day 365 |  | 15.3 [8.2 to 26.5] | 15.5 [8.4 to 26.9] | 3.2 [0.6 to 16.2]
  ST3 Day 29 |  | 6.9 [2.7 to 16.4] | 0.0 [0.0 to 6.2] | 3.1 [0.6 to 15.7]
  ST3 Day 57 |  | 77.6 [65.3 to 86.4] | 81.0 [69.1 to 89.1] | 3.0 [0.5 to 15.3]
  ST3 Day 85 |  | 94.9 [86.1 to 98.3] | 93.0 [83.3 to 97.2] | 3.0 [0.5 to 15.3]
  ST3 Day 180 |  | 74.1 [61.6 to 83.7] | 66.7 [53.7 to 77.5] | 6.3 [1.7 to 20.1]
  ST3 Day 236 |  | 38.2 [23.9 to 55.0] | 37.1 [23.2 to 53.7] | 5.6 [1.0 to 25.8]
  ST3 Day 365 |  | 13.6 [7.0 to 24.5] | 15.5 [8.4 to 26.9] | 3.2 [0.6 to 16.2]
  ST4 Day 29 |  | 3.4 [1.0 to 11.7] | 3.4 [1.0 to 11.7] | 0.0 [0.0 to 10.7]
  ST4 Day 57 |  | 55.2 [42.5 to 67.3] | 56.9 [44.1 to 68.8] | 0.0 [0.0 to 10.4]
  ST4 Day 85 |  | 89.8 [79.5 to 95.3] | 91.2 [81.1 to 96.2] | 0.0 [0.0 to 10.4]
  ST4 Day 180 |  | 55.2 [42.5 to 67.3] | 52.6 [39.9 to 65.0] | 0.0 [0.0 to 10.7]
  ST4 Day 236 |  | 29.4 [16.8 to 46.2] | 25.7 [14.2 to 42.1] | 5.6 [1.0 to 25.8]
  ST4 Day 365 |  | 16.9 [9.5 to 28.5] | 13.8 [7.2 to 24.9] | 6.5 [1.8 to 20.7]
  ST5 Day 29 |  | 3.4 [1.0 to 11.7] | 1.7 [0.3 to 9.1] | 0.0 [0.0 to 10.7]
  ST5 Day 57 |  | 55.2 [42.5 to 67.3] | 55.2 [42.5 to 67.3] | 0.0 [0.0 to 10.4]
  ST5 Day 85 |  | 84.7 [73.5 to 91.8] | 87.7 [76.8 to 93.9] | 0.0 [0.0 to 10.4]
  ST5 Day 180 |  | 51.7 [39.2 to 64.1] | 45.6 [33.4 to 58.4] | 3.1 [0.6 to 15.7]
  ST5 Day 236 |  | 29.4 [16.8 to 46.2] | 31.4 [18.6 to 48.0] | 5.6 [1.0 to 25.8]
  ST5 Day 365 |  | 8.5 [3.7 to 18.4] | 8.6 [3.7 to 18.6] | 3.2 [0.6 to 16.2]
  ST6 Day 29 |  | 5.2 [1.8 to 14.1] | 5.2 [1.8 to 14.1] | 0.0 [0.0 to 10.7]
  ST6 Day 57 |  | 51.7 [39.2 to 64.1] | 51.7 [39.2 to 64.1] | 0.0 [0.0 to 10.4]
  ST6 Day 85 |  | 88.1 [77.5 to 94.1] | 89.5 [78.9 to 95.1] | 0.0 [0.0 to 10.4]
  ST6 Day 180 |  | 53.4 [40.8 to 65.7] | 52.6 [39.9 to 65.0] | 6.3 [1.7 to 20.1]
  ST6 Day 236 |  | 26.5 [14.6 to 43.1] | 28.6 [16.3 to 45.1] | 5.6 [1.0 to 25.8]
  ST6 Day 365 |  | 15.3 [8.2 to 26.5] | 8.6 [3.7 to 18.6] | 3.2 [0.6 to 16.2]

9. Secondary Outcome: GMFRs (Geometric Mean of the Fold Rise as Compared to Baseline) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 18 - 49 Years
Description: GMFRs (Geometric Mean of the Fold Rise as Compared to Baseline) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6), stratified by age group - Group 18 - 49 years.
  Calculations are based on number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean of the Fold Rise
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 133 | 136 | 88
Geometric Mean of the Fold Rise
  ST1 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST1 Day 57 | 1.6 [1.2 to 2.1] | 1.7 [1.5 to 2.0] | 2.2 [1.8 to 2.6] | 1.0 [1.0 to 1.1]
  ST1 Day 85 | 3.6 [2.2 to 5.6] | 5.3 [4.4 to 6.2] | 6.4 [5.3 to 7.7] | 1.0 [1.0 to 1.0]
  ST1 Day 180 | 1.3 [1.0 to 1.6] | 1.6 [1.4 to 1.8] | 1.7 [1.5 to 2.0] | 1.0 [1.0 to 1.0]
  ST1 Day 236 | 1.1 [0.9 to 1.3] | 1.3 [1.1 to 1.4] | 1.3 [1.1 to 1.6] | 1.0 [1.0 to 1.1]
  ST1 Day 365 | 1.0 [0.9 to 1.1] | 1.1 [1.1 to 1.2] | 1.2 [1.1 to 1.3] | 1.0 [1.0 to 1.1]
  ST2 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST2 Day 57 | 3.2 [2.2 to 4.7] | 4.5 [3.7 to 5.4] | 6.0 [5.1 to 7.2] | 1.0 [1.0 to 1.1]
  ST2 Day 85 | 8.4 [5.7 to 12.4] | 14.8 [12.9 to 17.0] | 16.0 [13.8 to 18.6] | 1.0 [1.0 to 1.0]
  ST2 Day 180 | 1.9 [1.4 to 2.7] | 3.2 [2.7 to 3.8] | 3.6 [3.0 to 4.2] | 1.0 [1.0 to 1.0]
  ST2 Day 236 | 1.2 [1.0 to 1.6] | 2.0 [1.7 to 2.3] | 1.8 [1.5 to 2.2] | 1.0 [1.0 to 1.0]
  ST2 Day 365 | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.4] | 1.0 [1.0 to 1.0]
  ST3 Day 29 | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST3 Day 57 | 5.0 [3.2 to 7.8] | 6.0 [5.0 to 7.3] | 7.9 [6.4 to 9.7] | 1.0 [1.0 to 1.1]
  ST3 Day 85 | 12.1 [8.6 to 17.0] | 14.7 [12.7 to 16.9] | 16.6 [14.0 to 19.6] | 1.0 [1.0 to 1.0]
  ST3 Day 180 | 2.4 [1.6 to 3.6] | 3.0 [2.6 to 3.5] | 3.6 [3.0 to 4.3] | 1.0 [1.0 to 1.0]
  ST3 Day 236 | 1.6 [1.2 to 2.2] | 1.8 [1.5 to 2.1] | 2.0 [1.6 to 2.4] | 1.0 [1.0 to 1.0]
  ST3 Day 365 | 1.2 [1.0 to 1.4] | 1.3 [1.2 to 1.4] | 1.4 [1.2 to 1.6] | 1.0 [1.0 to 1.0]
  ST4 Day 29 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST4 Day 57 | 2.1 [1.5 to 3.0] | 2.7 [2.3 to 3.2] | 3.5 [2.9 to 4.2] | 1.0 [1.0 to 1.0]
  ST4 Day 85 | 5.4 [3.5 to 8.5] | 8.6 [7.5 to 9.8] | 10.2 [8.6 to 12.0] | 1.0 [1.0 to 1.0]
  ST4 Day 180 | 1.5 [1.1 to 2.1] | 2.3 [2.0 to 2.7] | 2.6 [2.2 to 3.1] | 1.0 [1.0 to 1.1]
  ST4 Day 236 | 1.2 [0.9 to 1.5] | 1.7 [1.4 to 2.0] | 1.7 [1.4 to 2.0] | 1.0 [1.0 to 1.0]
  ST4 Day 365 | 1.1 [1.0 to 1.2] | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.0]
  ST5 Day 29 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 57 | 2.1 [1.5 to 3.0] | 2.8 [2.4 to 3.3] | 4.0 [3.3 to 4.8] | 1.0 [1.0 to 1.0]
  ST5 Day 85 | 5.7 [3.8 to 8.7] | 9.0 [7.8 to 10.3] | 10.8 [9.1 to 12.8] | 1.0 [1.0 to 1.0]
  ST5 Day 180 | 1.3 [1.0 to 1.7] | 2.1 [1.8 to 2.4] | 2.7 [2.3 to 3.2] | 1.0 [1.0 to 1.0]
  ST5 Day 236 | 1.1 [0.9 to 1.3] | 1.6 [1.4 to 1.8] | 1.6 [1.4 to 2.0] | 1.0 [1.0 to 1.0]
  ST5 Day 365 | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.3] | 1.3 [1.1 to 1.4] | 1.0 [1.0 to 1.0]
  ST6 Day 29 | 1.0 [1.0 to 1.0] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST6 Day 57 | 2.0 [1.4 to 2.8] | 2.6 [2.2 to 3.1] | 3.4 [2.8 to 4.2] | 1.0 [1.0 to 1.1]
  ST6 Day 85 | 5.4 [3.6 to 8.3] | 9.1 [7.9 to 10.4] | 10.6 [9.0 to 12.5] | 1.0 [1.0 to 1.0]
  ST6 Day 180 | 1.4 [1.1 to 1.9] | 2.3 [2.0 to 2.6] | 2.5 [2.2 to 3.0] | 1.0 [1.0 to 1.0]
  ST6 Day 236 | 1.2 [1.0 to 1.5] | 1.7 [1.5 to 2.0] | 1.7 [1.4 to 2.0] | 1.0 [1.0 to 1.1]
  ST6 Day 365 | 1.1 [1.0 to 1.3] | 1.2 [1.1 to 1.4] | 1.3 [1.2 to 1.5] | 1.0 [1.0 to 1.1]

10. Secondary Outcome: GMFRs (Geometric Mean of the Fold Rise as Compared to Baseline) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6) - Group 50 - 65 Years
Description: GMFRs (Geometric Mean of the Fold Rise as Compared to Baseline) for IgG (Immunoglobulin G) Against Each OspA (Outer Surface Protein A) Serotype (ST1 to ST6), stratified by age group - Group 50 - 65 years.
  Calculations are based on number of subjects with non-missing results.
Time Frame: up to Day 365 / Month 12
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean of the Fold Rise
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 0 | 59 | 58 | 33
Geometric Mean of the Fold Rise
  ST1 Day 29 |  | 1.2 [1.0 to 1.4] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1]
  ST1 Day 57 |  | 2.1 [1.6 to 2.8] | 1.8 [1.4 to 2.3] | 1.0 [0.9 to 1.1]
  ST1 Day 85 |  | 4.5 [3.3 to 6.1] | 4.5 [3.3 to 6.0] | 1.0 [1.0 to 1.1]
  ST1 Day 180 |  | 1.7 [1.4 to 2.1] | 1.6 [1.3 to 1.9] | 1.0 [1.0 to 1.1]
  ST1 Day 236 |  | 1.2 [1.0 to 1.5] | 1.3 [1.1 to 1.5] | 1.0 [1.0 to 1.1]
  ST1 Day 365 |  | 1.2 [1.0 to 1.3] | 1.1 [1.0 to 1.2] | 1.0 [0.9 to 1.1]
  ST2 Day 29 |  | 1.1 [0.9 to 1.3] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.1]
  ST2 Day 57 |  | 4.4 [3.2 to 6.1] | 4.1 [3.0 to 5.5] | 1.0 [1.0 to 1.1]
  ST2 Day 85 |  | 12.3 [9.5 to 15.8] | 13.3 [10.2 to 17.2] | 1.0 [1.0 to 1.1]
  ST2 Day 180 |  | 2.9 [2.3 to 3.8] | 2.9 [2.2 to 3.7] | 1.0 [1.0 to 1.1]
  ST2 Day 236 |  | 1.5 [1.2 to 1.9] | 1.6 [1.2 to 2.2] | 1.0 [1.0 to 1.0]
  ST2 Day 365 |  | 1.2 [1.1 to 1.5] | 1.2 [1.1 to 1.4] | 1.0 [1.0 to 1.1]
  ST3 Day 29 |  | 1.1 [1.0 to 1.4] | 1.0 [1.0 to 1.0] | 1.1 [0.9 to 1.2]
  ST3 Day 57 |  | 6.1 [4.3 to 8.7] | 5.9 [4.3 to 8.2] | 1.1 [0.9 to 1.2]
  ST3 Day 85 |  | 12.5 [9.6 to 16.4] | 12.8 [9.7 to 17.0] | 1.1 [0.9 to 1.2]
  ST3 Day 180 |  | 3.3 [2.6 to 4.2] | 3.0 [2.3 to 3.8] | 1.1 [1.0 to 1.2]
  ST3 Day 236 |  | 1.7 [1.3 to 2.2] | 1.8 [1.4 to 2.5] | 1.1 [0.9 to 1.3]
  ST3 Day 365 |  | 1.3 [1.1 to 1.5] | 1.2 [1.1 to 1.4] | 1.1 [0.9 to 1.2]
  ST4 Day 29 |  | 1.1 [0.9 to 1.3] | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST4 Day 57 |  | 2.7 [2.0 to 3.7] | 2.6 [2.0 to 3.3] | 1.0 [1.0 to 1.0]
  ST4 Day 85 |  | 7.4 [5.7 to 9.7] | 7.9 [6.1 to 10.2] | 1.0 [1.0 to 1.0]
  ST4 Day 180 |  | 2.2 [1.8 to 2.8] | 2.1 [1.7 to 2.5] | 1.0 [1.0 to 1.0]
  ST4 Day 236 |  | 1.4 [1.2 to 1.7] | 1.4 [1.1 to 1.7] | 1.1 [0.9 to 1.2]
  ST4 Day 365 |  | 1.2 [1.0 to 1.4] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.2]
  ST5 Day 29 |  | 1.1 [0.9 to 1.2] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  ST5 Day 57 |  | 2.9 [2.1 to 3.8] | 2.8 [2.1 to 3.6] | 1.0 [1.0 to 1.0]
  ST5 Day 85 |  | 7.8 [5.9 to 10.3] | 8.1 [6.2 to 10.6] | 1.0 [1.0 to 1.0]
  ST5 Day 180 |  | 2.2 [1.8 to 2.8] | 2.0 [1.6 to 2.6] | 1.0 [1.0 to 1.1]
  ST5 Day 236 |  | 1.4 [1.2 to 1.8] | 1.5 [1.2 to 1.9] | 1.1 [0.9 to 1.2]
  ST5 Day 365 |  | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.1]
  ST6 Day 29 |  | 1.1 [0.9 to 1.2] | 1.1 [1.0 to 1.2] | 1.0 [1.0 to 1.0]
  ST6 Day 57 |  | 2.6 [1.9 to 3.4] | 2.6 [2.0 to 3.4] | 1.0 [1.0 to 1.0]
  ST6 Day 85 |  | 7.9 [6.1 to 10.4] | 8.7 [6.7 to 11.3] | 1.0 [1.0 to 1.0]
  ST6 Day 180 |  | 2.3 [1.9 to 2.9] | 2.3 [1.8 to 2.9] | 1.1 [1.0 to 1.2]
  ST6 Day 236 |  | 1.4 [1.1 to 1.7] | 1.5 [1.2 to 1.9] | 1.1 [0.9 to 1.3]
  ST6 Day 365 |  | 1.2 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.2]

11. Secondary Outcome: Percentage of Participants With SAEs (Serious Adverse Events)
Description: Frequency of SAEs (Serious Adverse Events) during the entire study; frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 0.0 [0.0 to 11.7] | 1.9 [0.7 to 4.7] | 2.4 [1.0 to 5.6] | 2.4 [0.8 to 6.9]

12. Secondary Outcome: Percentage of Participants With Related SAEs (Serious Adverse Events)
Description: Frequency of related SAEs (Serious Adverse Events) during the entire study; frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 0.0 [0.0 to 11.7] | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 3.0]

13. Secondary Outcome: Percentage of Participants With AESIs (Adverse Events of Special Interest)
Description: Frequency of AESIs (Adverse Events of Special Interest) during the entire study; frequency is being assessed in terms of percentage of participants.
  AESIs are cases of Lyme Diseases, Lyme associated Events and the onset of potentially autoimmune or neuro-inflammatory disorders.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 0.0 [0.0 to 11.7] | 1.9 [0.7 to 4.7] | 0.5 [0.1 to 2.7] | 0.0 [0.0 to 3.0]

14. Secondary Outcome: Percentage of Participants With Related AESIs (Adverse Events of Special Interest)
Description: Frequency of related AESIs (Adverse Events of Special Interest) during the entire study; frequency is being assessed in terms of percentage of participants.
  AESIs are cases of Lyme Diseases, Lyme associated Events and the onset of potentially autoimmune or neuro-inflammatory disorders.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 0.0 [0.0 to 11.7] | 0.5 [0.1 to 2.6] | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 3.0]

15. Secondary Outcome: Percentage of Participants With Unsolicited AEs (Adverse Events)
Description: Frequency of unsolicited AEs (Adverse Events) during the entire study (incl. clinically relevant laboratory parameters); frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 27.6 [14.7 to 45.7] | 51.9 [45.2 to 58.5] | 56.6 [49.7 to 63.2] | 51.6 [42.9 to 60.2]

16. Secondary Outcome: Percentage of Participants With Related Unsolicited AEs (Adverse Events)
Description: Frequency of related unsolicited AEs (Adverse Events) during the entire study (incl. clinically relevant laboratory parameters); frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants | 6.9 [1.9 to 22.0] | 9.3 [6.1 to 14.0] | 14.6 [10.4 to 20.1] | 8.9 [5.0 to 15.2]

17. Secondary Outcome: Percentage of Participants With Solicited Local and Solicited Systemic AEs (Adverse Events)
Description: Frequency of solicited local and solicited systemic AEs (Adverse Events) within 7 days after each and after any vaccination; frequency is being assessed in terms of percentage of participants.
Time Frame: Day 1 (day of first vaccination) through Day 7; Day 29 (day of second vaccination) through Day 35; Day 57 (day of third vaccination) through Day 63
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
percentage of participants
  Solicted Local AEs | 89.7 [73.6 to 96.4] | 93.0 [88.8 to 95.7] | 96.1 [92.5 to 98.0] | 29.8 [22.5 to 38.4]
  Solicited Systemic AEs | 62.1 [44.0 to 77.3] | 67.8 [61.2 to 73.7] | 71.7 [65.2 to 77.4] | 42.7 [34.4 to 51.5]

18. Secondary Outcome: Percentage of Participants With SAEs (Serious Adverse Events), AESIs (Adverse Events of Special Interest), Solicited and Unsolicited AEs (Adverse Events) - Group 18-49
Description: Frequency of SAEs (Serious Adverse Events), AESIs (Adverse Events of Special Interest), solicited and unsolicited AEs (Adverse Events) during the entire study stratified by age group - Group 18-49; frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Population: The overall number analyzed is for all participants. Below listed number of participants is for the different age groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 147 | 145 | 91
percentage of participants
  SAEs | 0.0 [0.0 to 11.7] | 2.0 [0.7 to 5.8] | 2.1 [0.7 to 5.9] | 1.1 [0.2 to 6.0]
  AESIs | 0.0 [0.0 to 11.7] | 0.7 [0.1 to 3.8] | 0.0 [0.0 to 2.6] | 0.0 [0.0 to 4.1]
  solicited AEs | 89.7 [73.6 to 96.4] | 93.9 [88.8 to 96.7] | 96.6 [92.2 to 98.5] | 56.0 [45.8 to 65.8]
  unsolicited AEs | 27.6 [14.7 to 45.7] | 49.0 [41.0 to 57.0] | 55.2 [47.0 to 63.0] | 50.5 [40.5 to 60.6]

19. Secondary Outcome: Percentage of Participants With SAEs (Serious Adverse Events), AESIs (Adverse Events of Special Interest), Solicited and Unsolicited AEs (Adverse Events) - Group 50-65 Years
Description: Frequency of SAEs (Serious Adverse Events), AESIs (Adverse Events of Special Interest), Solicited and Unsolicited AEs (Adverse Events) during the entire study stratified by age group - Group 50-65 years; frequency is being assessed in terms of percentage of participants.
Time Frame: up to Day 365 / Month 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 0 | 67 | 60 | 33
percentage of participants
  SAEs |  | 1.5 [0.3 to 8.0] | 3.3 [0.9 to 11.4] | 6.1 [1.7 to 19.6]
  AESIs |  | 4.5 [1.5 to 12.4] | 1.7 [0.3 to 8.9] | 0.0 [0.0 to 10.4]
  solicited AEs |  | 92.5 [83.7 to 96.8] | 96.7 [88.6 to 99.1] | 51.5 [35.2 to 67.5]
  unsolicited AEs |  | 58.2 [46.3 to 69.3] | 60.0 [47.4 to 71.4] | 54.5 [38.0 to 70.2]

20. Secondary Outcome: Number of Participants With AESIs (Adverse Events of Special Interest) up to Study End
Time Frame: up to Day 365 / Month 12
Measure: Number; unit: Number of participants
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
Number analyzed (Participants) | 29 | 214 | 205 | 124
Number of participants
  Any AE of Special Interest | 0 | 4 | 1 | 0.
  Lyme disease | 0 | 2 | 0 | 0
  Erythema migrans | 0 | 1 | 0 | 0
  Osteoarthritis | 0 | 1 | 0 | 0
  Polyarthritis | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: up to Day 365
Description: Solicited AEs comprised injection site reactions (pain, itching, tenderness, induration (hardening), swelling, erythema (redness)) or systemic reactions (headache, muscle pain, fever (oral), flu-like symptoms, nausea, vomiting, rash, excessive fatigue). Solicited AEs are collected by systematic assessment through subject diaries (up to 7 days after each vaccination) and unsolicited AEs, SAEs and AESIs are collected through non-systematic assessment up to Day 365.
Arm/Group | VLA15 Low Dose | VLA15 Medium Dose | VLA15 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/214 | 0/205 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/29 | 4/214 | 5/205 | 3/124
Other Adverse Events (participants affected / at risk) | 26/29 | 203/214 | 202/205 | 85/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA15 Low Dose (N=29) | VLA15 Medium Dose (N=214) | VLA15 High Dose (N=205) | Placebo (N=124)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA15 Low Dose (N=29) | VLA15 Medium Dose (N=214) | VLA15 High Dose (N=205) | Placebo (N=124)
Injection site pain (General disorders) | 26 (111) | 198 (924) | 196 (941) | 30 (57) — includes systematic and non-systematic assessments
Fatigue (General disorders) | 8 (14) | 66 (111) | 81 (130) | 29 (40) — includes systematic and non-systematic assessments
Injection site erythema (General disorders) | 8 (10) | 68 (116) | 72 (123) | 12 (18)
Injection site induration (General disorders) | 3 (6) | 64 (108) | 65 (108) | 2 (3)
Injection site swelling (General disorders) | 4 (6) | 57 (84) | 68 (104) | 4 (6)
Influenza like illness (General disorders) | 3 (3) | 32 (44) | 42 (49) | 20 (25) — includes systematic and non-systematic assessments
Pyrexia (General disorders) | 2 (2) | 9 (10) | 7 (7) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (22) | 106 (173) | 97 (156) | 21 (29) — includes systematic and non-systematic assessments
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 42 (67) | 37 (55) | 12 (23) — includes systematic and non-systematic assessments
Headache (Nervous system disorders) | 10 (19) | 73 (115) | 84 (135) | 33 (46) — includes systematic and non-systematic assessments
Nausea (Gastrointestinal disorders) | 5 (5) | 23 (31) | 32 (36) | 11 (15)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 14 (16) | 10 (12) | 7 (8)
Nasopharyngitis (Infections and infestations) | 0 (0) | 9 (10) | 10 (11) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03769194/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT03769194/SAP_001.pdf